CLINICAL TRIAL: NCT02012803
Title: Conservative vs. Operative Treatment of Achilles Tendon Rupture, Prospective Randomized Controlled Trial
Brief Title: Achilles Tendon Rupture, Conservative vs. Operative Treatment: Prospective Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Evo-rad-akilles-2
Record Dates: First submitted 2013-11-27; First posted 2013-12-16 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture; treatment, elongation; operative treatment of achilles tendon rupture; conservative treatment of achilles tendon rupture

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative treatment (Experimental)
  Interventions: Procedure: End to end suturation by Krackow locking loop surgical technique with 2-Fiber-Wire suture
- conservative treatment (Active Comparator)
  Interventions: Other: Conservative treatment of achilles tendon rupture

INTERVENTIONS:
Procedure: End to end suturation by Krackow locking loop surgical technique with 2-Fiber-Wire suture — Operative treatment of achilles tendon rupture; End to end suturation by Krackow locking loop surgical technique with 2-Fiber-Wire suture and after operation identical protocol as conservative treatment.
  Arms: Operative treatment
Other: Conservative treatment of achilles tendon rupture — Conservative treatment of achilles tendon rupture; 1 week equinus-cast without bearing, and then 6 week Vacoped orthosis with different equinus degrees and full weight bearing.
  Arms: conservative treatment

SUMMARY:
The intention is to compare prospectively operative and conservative early functional rehabilitation protocol in treatment of total achilles tendon rupture. To compare these treatments, the investigators use 1998 published Leppilahti-score, Rand-36 quality of life-questionnaire and MRI. The Leppilahti-score includes both subjective and objective items (pain, stiffness, subjective calf muscle weakness, footwear restrictions, active range of motion between ankles, subjective result, isokinetic calf muscle strength). The investigators also study MRI-imaging for both legs and compare including achilles tendon elongation and muscle volume correlations to Leppilahti-score results between these two treatments. Follow-up time is 18 months.

Hypothesis is that operative treatment offers no benefit in comparison conservative treatment, with identical rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years, Clinical diagnosis of total achilles tendon rupture, ultrasonography controlled tendon ends reposition when ankle is in equinus/ plantar flexion.

Exclusion Criteria:

* earlier achilles tendon disorders, corticosteroid injections in achilles tendon, fluorokinolol-antibiotics in 2 years earlier, systemic corticosteroid medication, diabetes, peripheral arterial disease, more than 7 days old rupture, patient lives abroad or patient refused to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Subjective and objective results in conservative and operative treatment of Achilles tendon rupture. | 18 months
  Subjective results consists of Rand-36 questionnaire and part of Leppilahti-scores questionnaire. Objective results consists of calf muscle isokinetic strength measurements and MRI-findings.

SECONDARY OUTCOMES:
Complications in treatment of achilles tendon rupture. | 18 months
  Complications are re-rupture and postoperative infection.
Achilles tendon MRI-findings in operative and conservative treatment of achilles tendon rupture. | 18 months
  We study calf muscle volume, achilles tendon volume, fat degeneration and achilles tendon elongation.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Heikkinen J, Lantto I, Flinkkila T, Ohtonen P, Niinimaki J, Siira P, Laine V, Leppilahti J. Soleus Atrophy Is Common After the Nonsurgical Treatment of Acute Achilles Tendon Ruptures: A Randomized Clinical Trial Comparing Surgical and Nonsurgical Functional Treatments. Am J Sports Med. 2017 May;45(6):1395-1404. doi: 10.1177/0363546517694610. Epub 2017 Mar 10. PMID 28282504
- [Derived] Lantto I, Heikkinen J, Flinkkila T, Ohtonen P, Siira P, Laine V, Leppilahti J. A Prospective Randomized Trial Comparing Surgical and Nonsurgical Treatments of Acute Achilles Tendon Ruptures. Am J Sports Med. 2016 Sep;44(9):2406-14. doi: 10.1177/0363546516651060. Epub 2016 Jun 15. PMID 27307495